CLINICAL TRIAL: NCT00226733
Title: Training Intensity After Coronary Bypass Grafting
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other); Landsforeningen for hjerte og lungesyke (LHL) (Unknown); Røros Rehabiliteringssenter (Unknown); St. Olavs Hospital (Other)
Responsible Party: Trine Moholdt, Norwegian University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BypassRoros1
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2008-04

CONDITIONS: Coronary Artery Bypass
Keywords: Coronary Artery Bypass (E04.928.220.520.220); Exercise Test [E01.370.370.380.250]; Echocardiography [E01.370.370.380.220]; Quality of Life [K01.752.400.750]
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Interval exercise training with high intensity
  Interventions: Behavioral: Exercise training
- B (Active Comparator): Exercise training with moderate intensity
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Interval exercise training with high intensity five days per week for four weeks.
  Arms: A
Behavioral: Exercise training — Exercise training with moderate intensity, five days per week for four weeks.
  Arms: B

SUMMARY:
The purpose of this study is to investigate the effect of high and moderate intensity exercise training after coronary bypass surgery. The subjects are randomised to training at either 60-70% or 85-95% of their maximal capacity daily for four weeks. Primary outcome measure is change in maximal aerobic capacity, measured as change in maximal oxygen consumption, after the training period. Secondary outcome measures are change in quality of life, heart rate variability, ultrasound measures of the heart and blood variables, including endothelian markers.

DETAILED DESCRIPTION:
The exercise part of cardiac rehabilitation today is often composed of low to moderate intensity training. Several studies have found interval training with high intensity to be more effective in improving physical capacity in healthy subjects and also in different patient populations. We therefore wish to compare high intensity interval training with moderate intensity training in patients operated with coronary bypass surgery. Maximal oxygen consumption is shown to be the best indicator of how many years you life, both in healthy persons and in cardiac patients.

The subjects in this study is attending a four week rehabilitation program at an residential institution in Norway. They are randomised to do either a moderate or a high intensity aerobic training session each day.

The hypothesis in advance, was that high intensity interval training lead to a greater improvement in maximal oxygen consumption than training with moderate intensity. We also hypothesised that there would be no difference between the two groups after 6 months, since then the patients had to administer their own exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Grafting (4-12 weeks ago)

Exclusion Criteria:

* Not able to exercise on a treadmill
* Left ventricle ejection fraction < 30%
* hemodynamic significant valve deficit (> NYHA classification II)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Oxygen Consumption

SECONDARY OUTCOMES:
Quality of life
Pulse
Blodverdier
Ekkokardiografiske parametre

CONTACTS AND LOCATIONS:
Overall Officials: Stig A Slørdahl, Dr.med, Study Chair — NTNU, Institutt for sirkulasjon og bildediagnostikk; Trine T Moholdt, MS, Principal Investigator — NTNU, Institutt for sirkulasjo og bildediagnostikk
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway